CLINICAL TRIAL: NCT05047042
Title: Advanced Cancer Support In Virtual Rehabilitation and Exercise in North Zone (ACTIVE-North): a Feasibility Study
Brief Title: A Feasibility Study of a Virtual Rehabilitation and Physical Activity Program for People With Advanced Cancer
Acronym: ACTIVE-North
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Alberta Health services (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HREBA.CC-21-0301
Record Dates: First submitted 2021-09-08; First posted 2021-09-16 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Advanced Cancer
Keywords: exercise; rehabilitation
MeSH Terms: conditions — Motor Activity | interventions — Telerehabilitation; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Advanced Cancer Support in Virtual Rehabilitation and Exercise (Experimental): The intervention will take place in participants' homes, at times convenient for the participant. Programming will be administered virtually through the University of Alberta's Cancer Rehabilitation Clinic, which is fully equipped for virtual delivery of services. The study intervention will be tailored to the individual with respect to their baseline strength, symptom profile and prior experience with exercise. Pre- and post-testing will be done virtually. The mode, intensity and duration of each exercise session will be based on the participant's baseline fitness and status that day. Variations on each exercise will be provided to ensure an appropriate movement and intensity and to allow for individual prescription. Resistance bands will be used to provide resistance during strengthening and balance retraining exercises. The interactive group class will be led virtually by an exercise or rehabilitation specialist.
  Interventions: Behavioral: Advanced Cancer Support in Virtual Rehabilitation and Exercise

INTERVENTIONS:
Behavioral: Advanced Cancer Support in Virtual Rehabilitation and Exercise — The study intervention will consist of an individualized 8-week program of online exercise modules, supervised interactive group class and one-to-one consultations with an exercise or rehabilitation specialist and a pain and symptom physician, delivered via secure live Zoom sessions.

SUMMARY:
Background: People with advanced cancer experience fatigue and loss of functioning, which often worsens as their cancer progresses. Rehabilitation programs may help to reduce fatigue and improve overall physical function. People with advanced cancer who live in rural and remote areas lack access to cancer-specific rehabilitation and exercise expertise to manage complex symptoms of high intensity. Their access to in-person services at tertiary sites are further reduced due to public health requirements for physical distancing during the severe acute respiratory syndrome coronavirus 2 pandemic. Aim: To test the feasibility of a virtual program delivered by a team of cancer-specific rehabilitation, exercise and pain and symptom experts for remote and rural patients with advanced cancer to address their symptoms, functioning and quality of life. Design: The virtual program will be tailored to the individual person, and consist of online exercise modules, online supervised interactive group class and one-to-one virtual meetings with an exercise or rehabilitation specialist and a palliative care physician. Relevance: This study will determine whether a virtual multidisciplinary rehabilitation and exercise program is feasible for people with advanced cancer. Further, it will provide insight on how fatigue and loss of functioning can best be managed for this population in remote and rural locations.

DETAILED DESCRIPTION:
Aim: To determine the feasibility of a virtual rehabilitation and therapeutic exercise intervention which is designed and delivered virtually by an interdisciplinary team for advanced cancer patients in Alberta Health Services North Zone. Objectives: 1) To examine the primary feasibility outcome of completion rate, with a target of 50% of participants who complete the virtual rehabilitation and therapeutic exercise intervention out of all participants who agreed to participate in the study; 2) To explore secondary feasibility outcomes of retention rate, adherence rate and patient safety of participants in the virtual rehabilitation and therapeutic exercise intervention; 3) To provide preliminary data on the effect of a virtual rehabilitation and therapeutic exercise intervention on the symptom burden, physical function, and overall quality of life of advanced cancer patients, and 4) To explore participants' experience, barriers, and facilitators after participating in the virtual rehabilitation and therapeutic exercise intervention. Methods: A pilot study using single group pre- to post-test with mixed methods data collection will allow us to determine the feasibility of a virtual rehabilitation and therapeutic exercise intervention (proof of concept) to be used in the full-scale study.

ELIGIBILITY:
Inclusion Criteria:

1. The ability to understand, provide informed consent in, and speak English;
2. Patient reported fatigue or loss of physical functioning of moderate to severe severity (Edmonton Symptom Assessment System - Revised score ≥ 4/10);
3. Primary residence in Alberta Health Services North Zone;
4. Internet access in the patient's home residence.

Exclusion Criteria:

1. Any absolute contraindications to exercise (including acute myocardial infarction within 2 days, symptomatic/severe aortic stenosis, decompensated heart failure, symptomatic/hemodynamically significant cardiac arrhythmias, unstable angina not previously stabilized by medical therapy, acute aortic dissection, acute myocarditis/pericarditis, acute pulmonary embolus/infarction);
2. Palliative Performance Scale level of 30% or less;
3. Any person who, in the opinion of the treating physician, is within the last days to hours of life.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2022-01-17 (Actual); Primary Completion 2024-02-05 (Actual); Study Completion 2024-02-05 (Actual)

PRIMARY OUTCOMES:
Completion rate | 12 months
  The number of participants who complete the study intervention, out of the total number of patients who agree to participate in the study intervention

SECONDARY OUTCOMES:
Retention rate | 12 months
  The number of participants completing the post-testing assessments, out of the total number of patients who agree to participate in the study intervention
Adherence rate | 12 months
  The number of sessions attended by the participant as a proportion of the maximum prescribed
Patient safety | 12 months
  The number and type of adverse events which may arise during the study intervention, including but limited to death, a life-threatening event, inpatient hospitalization, or a persistent or significant incapacity or substantial disruption of the ability to conduct basic activities of daily living.

OTHER OUTCOMES:
Patient-reported symptom severity | 8 weeks
  Edmonton Symptom Assessment System - Revised: Symptom severity or intensity is rated on an 11-point scale (0 = no symptom, 10 = worst possible symptom), with higher scores indicating worse symptom intensity.
Patient-reported fatigue | 8 weeks
  Brief Fatigue Inventory: Patient-rated numerical scale comprised of 9 items; the first three items ask patients to rate the severity of their fatigue at its "worst," "usual," and "now" during normal waking hours, with 0 being "no fatigue" and 10 being "fatigue as bad as you can imagine." The last six items assess the amount that fatigue has interfered with different aspects of the patient's life during the past 24 hours.
Patient-reported lower extremity functioning | 8 weeks
  Lower Extremity Functional Scale: Patient questionnaire administered by the study coordinator and comprised of 20 items; each item is an activity rated on a 5-point scale (0 = extreme difficulty or unable to perform activity, 4 = no difficulty).
Patient-reported upper extremity functioning | 8 weeks
  Upper Extremity Functional Scale: Patient questionnaire comprised of 8 items; each item is an activity rated on a 10-point scale (1 = no problem, 10 = major problem / can't do at all).
Objective functional lower extremity strength | 8 weeks
  Sit to Stand Test
Objective functional flexibility of lower back and hamstring muscles | 8 weeks
  Sit and Reach Test
Objective shoulder range of motion | 8 weeks
  Shoulder range of motion
Objective measure of static balance | 8 weeks
  4-stage balance test
Objective measure of aerobic and lower body endurance | 8 weeks
  2-minute step test

CONTACTS AND LOCATIONS:
Overall Officials: Margaret McNeely, PhD, Principal Investigator — University of Alberta, Faculty of Rehabilitation Medicine; Sonya Lowe, MD PhD, Principal Investigator — University of Alberta, Department of Oncology
Locations (3):
- Canada (3):
  - Cross Cancer Institute, Edmonton, Alberta
  - Fort McMurray Community Cancer Centre, Fort McMurray, Alberta
  - Grande Prairie Regional Cancer Centre, Grande Prairie, Alberta